CLINICAL TRIAL: NCT00133874
Title: An Observer-blind, Multicenter, Non-inferiority, Comparative Study of the Safety and Efficacy of Topical 1% SB-275833 Ointment, Applied Twice Daily for 5 Days, Versus Topical 2% Fusidic Acid Cream Applied Three Times Daily for 7 Days in the Treatment Adult and Paediatric Subjects With Impetigo
Brief Title: Topical SB-275833 Ointment, 1% For The Treatment Of Impetigo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TOC100224
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Skin Infections, Bacterial
Keywords: topical antibacterial; topical antibiotic; impetigo
MeSH Terms: conditions — Cellulitis; Impetigo

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB-275833 ointment, 1%
  Other Names: SB-275833 ointment; 1%

SUMMARY:
The goal of this study is to determine if topical SB-275833 ointment, 1% is as safe and effective as topical sodium fusidate ointment, 2% for the treatment of impetigo in adults and children as young as 9 months of age.

DETAILED DESCRIPTION:
A Randomised, Observer-blind, Multicentre, Non-inferiority, Comparative, Phase III Study of the Safety and Efficacy of Topical 1% SB-275833 Ointment, Applied Twice Daily for 5 Days, versus Topical 2% Sodium Fusidate Ointment Applied Three Times Daily for 7 Days in the Treatment of Adult and Paediatric Subjects with Impetigo.

ELIGIBILITY:
Inclusion criteria:

* Must have primary impetigo with total lesion area being 100 square centimeters or less.
* Women who could bear children must have a negative urine pregnancy test and agree to either abstain from sexual intercourse or the use of specific effective contraceptive measures.

Exclusion Criteria:

* Any signs and symptoms of systemic infection.
* Any serious underlying disease that could be imminently life threatening.

Min Age: 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2005-04; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Clinical response assessed at end of therapy visit. Clinical success defined by the need for no additional antibiotic treatment. | 7 Days

SECONDARY OUTCOMES:
Clinical response assessed at follow up visit. Microbiologic response at end of therapy and follow up visits. Impetigo lesion area measured at end of therapy and follow up visits. | 7 Days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (64):
- Canada (6):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, Toronto, Ontario
- GSK Investigational Site, San José, Costa Rica
- France (7):
  - GSK Investigational Site, Anzin
  - GSK Investigational Site, Bersée
  - GSK Investigational Site, Labarth-Sur-Leze
  - GSK Investigational Site, Martigues
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Seraincourt
  - GSK Investigational Site, Vieux-Condé
- Germany (25):
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Gilching, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Mahlow, Brandenburg
  - GSK Investigational Site, Duelmen, Lower Saxony
  - GSK Investigational Site, Bad Honnef, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Gelsenkirchen, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Mülheim, North Rhine-Westphalia
  - GSK Investigational Site, Olpe, North Rhine-Westphalia
  - GSK Investigational Site, Unna, North Rhine-Westphalia
  - GSK Investigational Site, Wuppertal, North Rhine-Westphalia
  - GSK Investigational Site, Worms, Rhineland-Palatinate
  - GSK Investigational Site, Döbeln, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Reichenbach, Saxony
  - GSK Investigational Site, Schmiedeberg, Saxony
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Preetz, Schleswig-Holstein
  - GSK Investigational Site, Rendsburg, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- India (2):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Mumbai
- Mexico (2):
  - GSK Investigational Site, Zapopan, Jalisco, Jalisco
  - GSK Investigational Site, Mexico City
- Netherlands (9):
  - GSK Investigational Site, Ermelo
  - GSK Investigational Site, Huizen
  - GSK Investigational Site, Losser
  - GSK Investigational Site, Musselkanaal
  - GSK Investigational Site, Oude Pekela
  - GSK Investigational Site, Sittard
  - GSK Investigational Site, Soerendonk
  - GSK Investigational Site, Zieuwent
  - GSK Investigational Site, Zwijndrecht
- GSK Investigational Site, Breña, Peru
- Poland (5):
  - GSK Investigational Site, Grudziądz
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Zabrze
- South Africa (6):
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Daveyton
  - GSK Investigational Site, Eloffsdal, Pretoria
  - GSK Investigational Site, Newtown
  - GSK Investigational Site, Pretoia
  - GSK Investigational Site, Pretoria

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: TOC100224 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: TOC100224 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: TOC100224 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: TOC100224 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: TOC100224 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: TOC100224 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: TOC100224 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register